CLINICAL TRIAL: NCT07112976
Title: Effect of a Higher Positive End-expiratory Pressure (PEEP) on Lung Hyperinflation and Collapse in Patients With Severe Pneumonia: a Computed Tomography Study
Brief Title: Lung Response to a Higher PEEP During Severe Pneumonia: a CT Study
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: Studio retrospettivo n. 28/25
Record Dates: First submitted 2025-07-03; First posted 2025-08-08 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Severe Pneumonia
Keywords: Mechanical ventilation; Positive end-expiratory pressure; Hyperinflation; Recruitment; Computed tomography
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
At their institution, the investigators routinely assess the individual response of mechanically ventilated patients with acute respiratory failure to higher positive end-expiratory pressure (PEEP) by examining changes in lung aeration through lung computed tomography (CT). They typically obtain two lung CT scans during an end-expiratory hold, one at a PEEP of 10 cmH2O and another at 15 cmH2O. Recruitment and hyperinflation are measured by assessing the decrease in the volume of non-aerated lung regions (with a density greater than -100 HU) and the increase in the volume of hyperinflated lung regions (with a density of less than -900 HU) between the two CT scans. If recruitment exceeds hyperinflation, the response to higher PEEP is considered "positive", and medical doctors are encouraged to treat that patient with a higher PEEP. Conversely, if hyperinflation exceeds recruitment, the response is deemed "negative", and a higher PEEP is discouraged. This assessment is further complemented by a "PEEP test," during which gas exchange (specifically arterial oxygen and carbon dioxide tension) and respiratory system mechanics (including compliance) are evaluated while ventilating with PEEP levels of 10 and 15 cmH2O.

In this retrospective analysis, the investigators will focus on patients with severe pneumonia who underwent the two lung CTs as part of their routine clinical practice. They will retrieve data on primary demographic characteristics, significant comorbidities, causes of pneumonia, severity of acute illness, and treatments delivered. Additionally, they will review the results of the quantitative analysis of the lung CT scans taken at 10 and 15 cmH2O, and the PEEP tests. The primary aim of this study is to determine the proportion of patients with net hyperinflation in response to higher PEEP.

ELIGIBILITY:
Inclusion Criteria:

* adult (≥18 years of age) patients
* admitted to ICU from 1/10/2022 to 31/12/2024
* with severe pneumonia
* treated with mechanical ventilation
* who underwent the two lung CTs at 10 and 15 cmH2O

Exclusion Criteria

* pneumothorax
* pneumomediastinum
* lung CT was obtained with contrast medium to rule out pulmonary embolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults admitted to the ICU with severe pneumonia, treated with mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Lung response to a higher PEEP | The effects of a higher PEEP will be assessed by comparing the CT scans taken at ICU admission, with a PEEP of 10 or 15 cmH2O, within the same subject. Usually, the interval between the two CT scans is a few minutes.
  The primary study objective is to evaluate the effects of higher PEEP with quantitative analysis of lung CT scans in patients with severe pneumonia. We hypothesize that 50% of these patients will exhibit more hyperinflation than recruitment.
  We measure recruitment and hyperinflation by assessing the change in the volume of non-aerated lung regions (with a density greater than -100 HU) and hyperinflated lung regions (with a density of less than -900 HU) between the two CT scans.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Humanitas Research Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Protti A, Santini A, Pennati F, Chiurazzi C, Cressoni M, Ferrari M, Iapichino GE, Carenzo L, Lanza E, Picardo G, Caironi P, Aliverti A, Cecconi M. Lung Response to a Higher Positive End-Expiratory Pressure in Mechanically Ventilated Patients With COVID-19. Chest. 2022 Apr;161(4):979-988. doi: 10.1016/j.chest.2021.10.012. Epub 2021 Oct 16. PMID 34666011